CLINICAL TRIAL: NCT05359003
Title: A Feasibility Study of a Step-goal Based Physical Activity Intervention in People With Epilepsy
Brief Title: Steps for Epilepsy
Acronym: StEpi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00084252; UL1TR001420 (NIH)
Record Dates: First submitted 2022-04-28; First posted 2022-05-03 (Actual); Results first posted 2025-10-31 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2024-03

CONDITIONS: Epilepsy
Keywords: physical activity; step goal; tele health
MeSH Terms: conditions — Epilepsy; Motor Activity

STUDY DESIGN:
Intervention Model Description: A randomized, controlled trial with a two-arm, parallel group design with a healthy living education control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Physical Activity Intervention (Experimental): Participants in this arm will undergo a 12-week physical activity program aimed to achieve the equivalent of 8,000 steps per day (56,000 weekly steps). Includes weekly meetings with a trained health coach.
  Interventions: Behavioral: 12-week Physical Activity Program
- Arm 2: Control (No Intervention): Participants randomized to the healthy living education control group will continue to undergo standard care for 12 weeks with a phone call from the coach every 2 weeks on topics of healthy living (topics include: keeping a seizure diary, sleep, medication adherence, stress, diet, emotional health)

INTERVENTIONS:
Behavioral: 12-week Physical Activity Program — Participants in this arm will undergo a 12-week physical activity program aimed to achieve the equivalent of 8,000 steps per day (56,000 weekly steps). Includes weekly meetings with a trained health coach.
  Arms: Arm 1: Physical Activity Intervention

SUMMARY:
The purpose of this research study is to evaluate the feasibility of a 12-week, telehealth delivered, step-goal based physical activity intervention in people with epilepsy. The study team will also evaluate the physical activity profiles of people with epilepsy both at rest and when engaged in physical activity and gather information on the effect of the intervention on epilepsy and epilepsy associated comorbidities.

DETAILED DESCRIPTION:
This is a randomized, controlled, pilot trial to assess the feasibility of a 12-week telehealth delivered, step-goal based physical activity intervention in people with epilepsy. This will be carried out using a 2-arm, parallel group design with a healthy living education control. Participants will undergo formal exercise testing to establish a baseline fitness level and safety of participation. They will wear Garmin activity tracker on their wrist throughout the study to track their steps. During a 4 week baseline period, we will gather data on baseline physical activity levels and seizure frequency. Participants will then be randomized to either the intervention group or a healthy living education control group. The intervention group will undergo a 12-week, telehealth delivered, step goal based physical activity intervention with a goal of ultimately achieving at least 8,000 steps per day. The intervention will utilize social cognitive theory to encourage lasting behavior changes and have weekly group coaching sessions with a trained health and behavior change provider. The control group will receive education every two weeks but will not be given a coaching plan. The study will evaluate adherence to the intervention, sustainability of the intervention over 12 weeks after the formal coaching program ends, and acceptability of the intervention. The study will also investigate the physical activity profile of people with epilepsy both at rest and when asked to participate in physical activity with a self-selected intensity and bout duration. The study will collect information on the effect of the intervention on seizures, mood, quality of life, sleep, fitness, and heart-rate variability, as well as other epilepsy relevant outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Focal or generalized epilepsy, as determined clinically by a WFBH epileptologist with no significant consideration of an alternative diagnosis
* Access to a smartphone with application capabilities
* Internet access or cellular data plan to attend virtual sessions
* Able to ambulate independently

Exclusion Criteria:

* Diagnosis of nonepileptic or psychogenic spells
* Seizures associated with falls with injury (such as atonic seizures)
* Medical conditions that would limit ability to participate in an exercise intervention including: Stage III or IV Congestive Heart Failure (CHF); End-stage Renal Disease; Severe dementia or significant cognitive impairment that precludes participation in the intervention or limits ability to follow the study protocol; Uncontrolled hypertension (HTN) defined as systolic blood pressure greater than 180 mmHg and diastolic blood pressure greater than 110 mmHg at rest; Severe arthritis, amputations, or orthopedic problems that limit ambulatory ability
* Currently pregnant or plan to become pregnant during the study period (16 weeks)
* An active Central Nervous System (CNS) infection, demyelinating disease, degenerative neurologic disease or any CNS disease deemed to be progressive during the course of the study that may confound the interpretation of the study results
* Any clinically significant psychiatric illness, psychological, or behavioral problems that would interfere with the subject's ability to participate in the study.
* Unwilling or unable to comply with all study visits and procedures
* Participants who have <75% complete days of seizure recording in the study diary or step data via the Garmin device will not be randomized.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Halley Alexander, MD, Principal Investigator — Wake Forest Health Sciences
Locations (1):
- Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During a 4-week baseline period, the participants will continue their usual activity but will wear the Garmin and ActivPAL 4 and keep a study diary. We will use this to assess their baseline PA profiles and seizure frequency and to screen for adherence with device and diary use, as participants who have <75% complete days of seizure recording or step data via the Garmin will not be randomized.
Period: Overall Study
Arm/Group | Arm 1: Physical Activity Intervention | Arm 2: Control
Started | 15 | 6
Completed | 14 | 3
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Physical Activity Intervention | Arm 2: Control | Total
Number analyzed (Participants) | 15 | 6 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (12.0) | 33.7 (7.66) | 36.41 (10.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 3 | 13
  Male | 5 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 6 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 12 | 5 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Who Achieve Their Assigned Step Goal - Adherence
Description: As measured by average daily steps via the Garmin device over the last 4 weeks of the intervention period.
Time Frame: Week 12 to Week 16
Population: Pre-specified to collect data and report results for Arm 1: Physical Activity Intervention only.
Measure: Number (95% Confidence Interval); unit: Proportion
Arm/Group | Arm 1: Physical Activity Intervention
Number analyzed (Participants) | 15
Proportion | 0.267 [0.076 to 0.581]

2. Primary Outcome: Proportion of Participants Who Achieve Their Assigned Step Goal - Sustainability
Description: As measured by average daily steps via the Garmin device over the last 4 weeks of the maintenance period, will be calculated and 95% binomial confidence intervals generated.
Time Frame: Week 24 to Week 28
Population: Pre-specified to collect data and report results for Arm 1: Physical Activity Intervention only.
Measure: Number (95% Confidence Interval); unit: Proportion
Arm/Group | Arm 1: Physical Activity Intervention
Number analyzed (Participants) | 14
Proportion | 0.143 [0.018 to 0.423]

3. Secondary Outcome: Time Spent Sedentary
Description: Time spent sedentary during the last week of baseline as measured by the Garmin watch.
Time Frame: Week 4
Measure: Mean (95% Confidence Interval); unit: avg minutes per week spent sedentary
Arm/Group | Arm 1: Physical Activity Intervention | Arm 2: Control
Number analyzed (Participants) | 14 | 6
avg minutes per week spent sedentary | 4790 [4388 to 5194] | 3356 [1265 to 5448]

4. Secondary Outcome: Time Spent in Light Intensity Activity
Description: Time spent in light intensity in the last week of baseline as measured by the Garmin watch.
Time Frame: Week 4
Measure: Mean (95% Confidence Interval); unit: avg minutes per week in light intensity
Arm/Group | Arm 1: Physical Activity Intervention | Arm 2: Control
Number analyzed (Participants) | 14 | 6
avg minutes per week in light intensity | 364 [267 to 461] | 297 [239 to 355]

5. Secondary Outcome: Time Spent in Moderate Intensity Activity
Description: Time spent in moderate intensity in the last week of baseline as measured by the Garmin watch.
Time Frame: Week 4
Measure: Mean (95% Confidence Interval); unit: avg minutes per week in moderate
Arm/Group | Arm 1: Physical Activity Intervention | Arm 2: Control
Number analyzed (Participants) | 14 | 6
avg minutes per week in moderate | 99.6 [42.4 to 157] | 45 [6.88 to 83.1]

6. Secondary Outcome: Time Spent in Vigorous Intensity Activity
Description: Time spent in vigorous intensity in the last week of baseline as measured by the Garmin watch.
Time Frame: Week 4
Measure: Mean (95% Confidence Interval); unit: avg minutes per week in vigorous
Arm/Group | Arm 1: Physical Activity Intervention | Arm 2: Control
Number analyzed (Participants) | 14 | 6
avg minutes per week in vigorous | 81.6 [18.6 to 145] | 40.8 [-17.8 to 99.4]

7. Secondary Outcome: Exit Survey
Description: The scale ranges from 4-20 with higher scores indicating greater satisfaction with the study.
Time Frame: Week 28
Population: For the Control Group: 3 dropouts participants did not complete the survey, and 1 participant only partially completed this form. Only 2 were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Physical Activity Intervention | Arm 2: Control
Number analyzed (Participants) | 14 | 2
score on a scale | 18.43 (1.95) | 17.50 (2.12)

8. Secondary Outcome: Exercise Satisfaction Survey- Proportion of Participants With a 4 or Higher Response
Description: We will use the question "How satisfied were you with the exercise intervention?" with scale of 1-5, 1=VERY UNSATISFIED, 2=UNSATISFIED, 3=NEUTRAL, 4=SATISFIED, 5=VERY SATISFIED. Higher numbers denotes better outcomes. We will calculate the proportion of subjects who answer 4 or above.
Time Frame: Week 16
Population: Pre-specified to collect data and report results for Arm 1: Physical Activity Intervention only. Only 13 participants were analyzed because 1 participant dropped out and 1 participant did not complete the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Physical Activity Intervention
Number analyzed (Participants) | 13
Participants | 9

9. Secondary Outcome: Time Spent Sedentary
Description: Time spent sedentary during the last week of intervention as measured by the Garmin watch.
Time Frame: Week 16
Measure: Mean (95% Confidence Interval); unit: avg minutes per week spent sedentary
Arm/Group | Arm 1: Physical Activity Intervention | Arm 2: Control
Number analyzed (Participants) | 14 | 2
avg minutes per week spent sedentary | 5608 [5146 to 6071] | 5344 [4699 to 5989]

10. Secondary Outcome: Time Spent Sedentary
Description: Time spent sedentary during the last week of maintenance as measured by the Garmin watch.
Time Frame: Week 28
Measure: Mean (95% Confidence Interval); unit: avg minutes per week spent sedentary
Arm/Group | Arm 1: Physical Activity Intervention | Arm 2: Control
Number analyzed (Participants) | 11 | 1
avg minutes per week spent sedentary | 4266 [2977 to 5556] | 5697 [NA to NA] — cannot calculate CI due to n=1

11. Secondary Outcome: Time Spent in Light Intensity Activity
Description: Time spent in light intensity in the last week of intervention as measured by the Garmin watch.
Time Frame: Week 16
Measure: Mean (95% Confidence Interval); unit: avg minutes per week in light intensity
Arm/Group | Arm 1: Physical Activity Intervention | Arm 2: Control
Number analyzed (Participants) | 14 | 2
avg minutes per week in light intensity | 374 [181 to 567] | 355 [50.2 to 659]

12. Secondary Outcome: Time Spent in Light Intensity Activity
Description: Time spent in light intensity in the last week of maintenance as measured by the Garmin watch.
Time Frame: Week 28
Measure: Mean (95% Confidence Interval); unit: avg minutes per week in light intensity
Arm/Group | Arm 1: Physical Activity Intervention | Arm 2: Control
Number analyzed (Participants) | 11 | 1
avg minutes per week in light intensity | 305 [109 to 501] | 742 [NA to NA] — cannot calculate CI due to n=1

13. Secondary Outcome: Time Spent in Moderate Intensity Activity
Description: Time spent in moderate intensity in the last week of intervention as measured by the Garmin watch.
Time Frame: Week 16
Measure: Mean (95% Confidence Interval); unit: avg minutes per week in moderate
Arm/Group | Arm 1: Physical Activity Intervention | Arm 2: Control
Number analyzed (Participants) | 14 | 2
avg minutes per week in moderate | 175 [-4.19 to 353] | 110 [68.8 to 151]

14. Secondary Outcome: Time Spent in Moderate Intensity Activity
Description: Time spent in moderate intensity in the last week of maintenance as measured by the Garmin watch.
Time Frame: Week 28
Measure: Mean (95% Confidence Interval); unit: avg minutes per week in moderate
Arm/Group | Arm 1: Physical Activity Intervention | Arm 2: Control
Number analyzed (Participants) | 11 | 1
avg minutes per week in moderate | 179 [36.3 to 322] | 141 [NA to NA] — cannot calculate CI due to n=1

15. Secondary Outcome: Time Spent in Vigorous Intensity Activity
Description: Time spent in vigorous intensity in the last week of intervention as measured by the Garmin watch.
Time Frame: Week 16
Measure: Mean (95% Confidence Interval); unit: avg minutes per week in vigorous
Arm/Group | Arm 1: Physical Activity Intervention | Arm 2: Control
Number analyzed (Participants) | 14 | 2
avg minutes per week in vigorous | 61.7 [13.9 to 110] | 156 [-18.9 to 332]

16. Secondary Outcome: Time Spent in Vigorous Intensity Activity
Description: Time spent in vigorous intensity in the last week of maintenance as measured by the Garmin watch.
Time Frame: Week 28
Measure: Mean (95% Confidence Interval); unit: avg minutes per week in vigorous
Arm/Group | Arm 1: Physical Activity Intervention | Arm 2: Control
Number analyzed (Participants) | 11 | 1
avg minutes per week in vigorous | 57.3 [17.8 to 96.7] | 160 [NA to NA] — cannot calculate CI due to n=1

ADVERSE EVENTS:
Time Frame: 7 months (Day 0 - Week 28)
Description: Adverse Events include worsening of seizure frequency, falls, and injuries. These will be recorded by the participant in their study diary, which will be returned electronically daily.
  All other adverse events will be collected at each study visit (visits 2-4) by asking "have you had any health problems since your last visit?"
Groups:
- Arm 1: Exercise Intervention: Participants in this arm will undergo a 12-week physical activity program aimed to achieve the equivalent of 8,000 steps per day (56,000 weekly steps).
  12-week physical activity program: Program aimed to achieve the equivalent of 8,000 steps per day (56,000 weekly steps). Includes weekly meetings with a trained health coach.
- Arm 2: Control: Participants randomized to the wait-list attention control group will continue to undergo standard care for 12 weeks.
Arm/Group | Arm 1: Exercise Intervention | Arm 2: Control
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/6
Serious Adverse Events (participants affected / at risk) | 4/15 | 1/6
Other Adverse Events (participants affected / at risk) | 11/15 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Exercise Intervention (N=15) | Arm 2: Control (N=6)
Fall with injury that required medical attention (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Dizziness that resulted in ER visit (Cardiac disorders) | 1 (1) | 0 (0)
Weakness that resulted in ER visit (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Planned admission for electrode implant placement (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Exercise Intervention (N=15) | Arm 2: Control (N=6)
Skin irritation at site of activity monitor (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Seizure with minor injury (not during exercise) (Nervous system disorders) | 2 (2) | 1 (3)
Dizziness and vomiting (General disorders) | 0 (0) | 1 (1)
Bumped into furniture (General disorders) | 2 (2) | 1 (2)
Seizure frequency increased (Nervous system disorders) | 1 (1) | 0 (0) — Seizure activity noted in the daily diary indicated an increase in seizures from baseline. Per protocol, temporal relationship with exercise was reviewed and not temporally related to exercise.
Depression episode (Psychiatric disorders) | 2 (2) | 0 (0)
Headache or migraine (Nervous system disorders) | 3 (3) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Kidney stone (Renal and urinary disorders) | 1 (1) | 0 (0)
Lipoma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Lupus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Minor fall (Injury, poisoning and procedural complications) | 6 (8) | 0 (0)
Strep throat (General disorders) | 1 (1) | 0 (0)
Seizure within 30 min of physical activity (Nervous system disorders) | 2 (4) | 0 (0)
Routine surgery to replace battery medical device (Surgical and medical procedures) | 1 (1) | 0 (0)
Seizure frequency increased (Nervous system disorders) | 1 (1) | 0 (0) — Self-reported an increase of seizures (two seizures in one day)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-21): https://cdn.clinicaltrials.gov/large-docs/03/NCT05359003/Prot_SAP_001.pdf
  • Informed Consent Form (2024-05-08): https://cdn.clinicaltrials.gov/large-docs/03/NCT05359003/ICF_000.pdf